CLINICAL TRIAL: NCT05644769
Title: The Chymase Angiotensin-(1-12) Axis in Hypertensive Disease
Brief Title: Chymase Angiotensin-(1-12) Axis In Hypertensive Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Trinity Hypertension & Metabolic Research Institute (Other)
Collaborators: Wake Forest University Health Sciences (Other)
Responsible Party: Principal Investigator, Henry Anthony Punzi, Medical Director, Trinity Hypertension & Metabolic Research Institute
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PMC-64-0010
Record Dates: First submitted 2022-11-22; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Determine the presence of the human sequence of Ang-(1-12) in plasma on no medications (Active Comparator): Determine the presence of the human sequence of Ang-(1-2) in the plasma of ten normal male and female hypertensive patients at baseline on no medications.
  Interventions: Other: Determine the presence of Human sequence Ang-(1-12) on no medication
- Determine the presence of human sequence of Ang-(1-12) on Lisinopril 40 mg every day (Active Comparator): Determine the presence of the human sequence of Ang-(1-12) in the plasma of 10 normal male and female hypertensive patients at baseline and after four weeks on Lisinopril 40 mg every day
  Interventions: Drug: Human sequence Ang-(1-12) on Lisinopril 40mg every day

INTERVENTIONS:
Other: Determine the presence of Human sequence Ang-(1-12) on no medication — Determine the presence of the human sequence of Ang-(1-12) in the plasma of ten normal male and female hypertensive patients on no medication.
  Arms: Determine the presence of the human sequence of Ang-(1-12) in plasma on no medications
Drug: Human sequence Ang-(1-12) on Lisinopril 40mg every day — Determine the presence of the human sequence of Ang-(1-12) in the plasma of 10 normal male and female hypertensive patients after four weeks on Lisinopril 40 mg every day.
  Arms: Determine the presence of human sequence of Ang-(1-12) on Lisinopril 40 mg every day

SUMMARY:
Determine the presence of the human sequence of Angiotensin-(1-12) in plasma of ten untreated hypertensive subjects and after 4 week with Lisinopril 40 mg every day. Determine the blood pressure reduction with Lisinopril 40mg.

DETAILED DESCRIPTION:
Determine the presence of the human sequence of Ang-(1-12) in the plasma of ten normal male and female hypertensive patients at baseline and after 4 weeks on Lisinopril 40mg every day. Measure concentrations of Ang-(1-12) in either spot urine collections from ten male and female hypertensive patients at baseline and after 4 weeks of Lisinopril 40mg every day.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of reading, comprehending the consent process and providing written informed consent to participate in the study
2. Subject willing to comply with all study visits/procedures and be available for the duration of the study
3. Male or female 40 years of age to 75 years of age
4. Male and female subjects naive to anti-hypertensive medications or receiving no anti-hypertensive medication for at least 6 months prior to visit 1
5. Stage I-II hypertension defined as a baseline mean seated cuff Diastolic blood pressure of equal/over 90 mm Hg and equal/less 109 mm Hg and/or Systolic blood pressure equal/over 140 mm Hg and equal/less 179 mm Hg on visit 1
6. Women may be enrolled if all three of the following criteria are met:

Have a negative urine pregnancy test at visit 1, for females of childbearing potential Are not breastfeeding Do not plan to become pregnant during the study And if one of the following three criteria is met Have had a hysterectomy or tubal ligation at least six months prior to signing the informed consent form Have been postmenopausal for at least one year Are of childbearing potential and will practice one of the following methods of birth control though out the study: oral, patch, injectable, or implantable hormone contraception, intrauterine device, diaphragm plus spermicide or female condom plus spermicide. Abstinence, partner's vasectomy are not acceptable methods of contraception

Exclusion Criteria:

-

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Presence of human sequence of Ang-(1-12) in plasma ten untreated essential hypertensive subjects at baseline | At baseline
  Determine the presence of the human sequence of Ang-(1-12) in plasma of ten untreated hypertensive subjects at baseline

SECONDARY OUTCOMES:
Presence of human sequence of Ang-(1-12) in plasma of ten subjects on four weeks of treatment on Lisinopril 40 mg every day | Four weeks
  Determine the presence of the human sequence of Ang-(1-12) in the plasma of ten normal male and female hypertensive patients after four weeks on Lisinopril 40 mg every day

CONTACTS AND LOCATIONS:
Overall Officials: Henry Punzi, MD, Principal Investigator — Trinity Hypertension & Metabolic Researach Institute
Locations (1):
- Punzi Medical Center, Carrollton, Texas, United States

IPD SHARING:
Plan to Share IPD: No